CLINICAL TRIAL: NCT04014478
Title: A Prospective, Multicenter, Self-Control Clinical Trial to Evaluate Safety and Efficacy of Endovascular Denervation in Treatment of Cancer Pain
Brief Title: A Clinical Trial to Evaluate Safety and Efficacy of Endovascualr Denervation in Treatment of Cancer Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Golden Leaf MedTec Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GL-CT-20161201
Record Dates: First submitted 2019-07-01; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: Liver Cancer; Pancreas Cancer; Stomach Cancer; Bile Duct Cancer
Keywords: Cancer； Pain
MeSH Terms: conditions — Liver Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Bile Duct Neoplasms; Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endovascular Denervation (Experimental)
  Interventions: Device: Endovascular Denervation

INTERVENTIONS:
Device: Endovascular Denervation — A radiofrequency ablation catheter will be placed in abdominal aorta. At least 6 sites will be ablated with settings of temerature at 60 degree centigrade and time at 120 seconds.

SUMMARY:
A prospective, multicenter, self-control clinical trial aim to enroll 110 patients suffered from upper abdominal (liver, pancreas, stomach, etc.) cancers . Patients who have taken at least one opioid drug for pain for two weeks and still have a VAS pain scale greater than 6 will receive endovascular denervation (EDN). They will be followed up for 3 months. The VAS scales, quantity of analgesics as represented by morphine equivalent and quality of life scores will be compared before and after EDN. Safety parameters such as arterial deformation, embolism, infection, liver and kidney functions will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with ages of 25 to 75;
* Clinically diagnosed as primary or secondary upper abdominal cancers (liver, pancreas, stomach, etc);
* Patients who have taken at least one opioid drug for pain for two weeks and still have VAS pain scale 》6;
* Expected lifetime 》4 months;
* Agrees to take part in the trial and signs the written, informed consent.

Exclusion Criteria:

* Women who are pregnant, or breast feeding, or having pregancy plan;
* Bleeding tendency or other coagulation related diseases;
* Acute or severe systemic infection;
* Past history of receving denervation procedure in aorta;
* No plans for surgical or interventional procedures in 3 months;
* History of stroke or TIA within 2 weeks;
* Acute coronary events within 2 weeks;
* Other conditions that deem unsuitable for the procedure, in the opinions of investigators.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale Changes over the time | Pre-treatment; 1, 3, 15, 30, 60, and 90 days after treatment.
  Pain scale is evaluated as Woodforde Visual Analig Scale (VAS) method. The scale is from 0 to 10, with 0 being no pain, and 10 being unbearable pain.

SECONDARY OUTCOMES:
Morphine Equivalent Changes over the time | Pre-treatment; 1, 3, 15, 30, 60, and 90 days after treatment.
  All analgesics used will be calculated to Morphine Equivalent using published conversion factors.
Quality of Life Score Changes over the time | Pre-treatment; 1, 3, 15, 30, 60, and 90 days after treatment.
  Qulaity of Life Scores are obtained using Functional Assessment of Cancer Theray-Generic Scale (FACT-G) (v 4.0) sale. The score is from 0 to 108, with 0 being no quality of life, and 108 being highest quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Study Chair — Zhongda Hospital; zhong-Min Wang, MD, Principal Investigator — Shanghai JiaoTong University Affiliated RuiJin Hospital; Jian Wang, MD, Principal Investigator — Beijing University Affiliated the First Hospital; Wen-Tao Li, MD, Principal Investigator — Fudan University Affiliated Cancer Hospital; Chuan-Sheng Zheng, MD, Principal Investigator — HuaZhong University of Science and Technology Affiliated Union Hospital; Wei-Fu Lv, MD, Principal Investigator — China University of Science and Technology Affiliated the First Hospital; Jun-Hui Sun, MD, Principal Investigator — Zhejiang University Affiliated the First Hospital; Hao Xu, MD, Principal Investigator — XuZhou Medical College Affiliated Hospital; Ming Huang, MD, Principal Investigator — Yunnan Cancer Hospital; Li-Gong Lu, MD, Principal Investigator — The People's Hospital of Zhuhai City; Jian-Song Ji, MD, Principal Investigator — The Central Hospital of Lishui City

IPD SHARING:
Plan to Share IPD: Yes